CLINICAL TRIAL: NCT02730442
Title: An Open Label Study in Healthy Volunteers to Evaluate the Potential for Drug/Drug Interactions Between F901318 and Fluconazole
Brief Title: Study of Potential for Interaction of Fluconazole With F901318
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Celerion Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F01318-01-05-15
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-04

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — olorofim; Antifungal Agents; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single dose F901318 with fluconazole (Experimental): AUC0-t for F901318 will be assessed before and after 5 days of treatment with fluconazole oral
  Interventions: Drug: F901318; Drug: Fluconazole

INTERVENTIONS:
Drug: F901318 — Administration of F901318 intravenously
  Other Names: Antifungal agent
Drug: Fluconazole — Oral administration
  Other Names: Antifungal agent

SUMMARY:
This will be an open label study in two parts. In the first part, F901318 (dose 2 mg/kg IV over 4 hours, Day 1) will be followed by F901318 (2 mg/kg IV over 4 hours) given on Day 8, after dosing with fluconazole 800 mg daily for 1 day (Day 4) and 400 mg daily orally for 4 days (Days 5 to 8). Up to twenty subjects will be included in two cohorts which will undergo the same dosing schedules of fluconazole and F901318 and undergo the same procedures. The first cohort will consist of 12 subjects studied in two groups of six subjects each. If there is clearly a difference in F901318 kinetics detectable before and after dosing with fluconazole in this first cohort, the second cohort will not be studied. If there is no clear difference, the second cohort will also be studied to give a final result. In this cohort, based on the pharmacokinetic findings in cohort 1, the dose of F901318 may be increased to up to 4 mg/kg to establish a dose suitable for phase 2 evaluation. PK sampling for plasma F901318 will continue from before the first dose up to and including 72 hours after dosing. PK sampling for fluconazole will continue from before the first dose and up to 72 hours after the fifth dose. A follow up visit will be conducted 7 +/- 2 days after discharge from the clinical unit following completion of blood sampling following the second dose of F901318 and the fifth dose of fluconazole.

The second part of the study will take place if no appreciable change in the pharmacokinetics of either F901318 or fluconazole has been observed in either the first or the second cohorts in the first part of the study. This second part will enrol 12 subjects. These subjects will receive fluconazole 800 mg daily for one day (Day 1) and 400 mg daily orally for 4 days (Days 2 to 5) in combination with F901318 which will be given in a dose of up to 4 mg/kg IV bid for one day (Day 1) followed by 7 doses of intravenous F901318 up to 2.5 mg/kg bid (Days 2 to 5). Pharmacokinetic profiles of F901318 and fluconazole will be obtained during dosing and over a 72-hour period following the final dose of both compounds.

DETAILED DESCRIPTION:
Part 1

Treatment Period (Day -1 to Day 11; visit 2):

Subjects will be admitted to the clinical unit in the afternoon of Day -1 and will remain on site until completion of the 72-hour post fluconazole and F901318 dose study-related procedures on Day 11. Admission procedures (Day -1) include a review of inclusion/exclusion criteria, weight, vital signs, test for drugs of abuse, alcohol and smoking and pregnancy where appropriate (must be negative), and a review of concomitant medication and adverse events. Blood (haematology, clinical chemistry and coagulation function) and urine (urinalysis) will be obtained for safety evaluations. Breakfast will be taken 30-60 minutes prior to dosing)

Days 1 - 4: F901318 (2 mg/kg IV for cohort 1 and up to 4 mg/kg IV for cohort 2) over 4 hours will be administered on Day 1. Blood samples for determination of plasma levels of F901318 will be collected predose and at the following time points up to 72 hours post-dose:

1, 2, 3, 4, 4.25, 4.5, 5, 6, 8, 10, 12, 16, 20, 24, 38, 48, 72 hours

Blood pressure, and pulse (lying and standing), and core temperature will be recorded at the following times on Day 1:

Prior to dosing, 1, 2, 4, 6, 8, 12 and 24 hours following dosing.

Twelve lead ECGs will be recorded prior to dosing and 1, 4, 8, 12 and 24 hours after dosing with F901318.

Telemetry will be set up 1 hour prior to dosing with F901318 and will continue for 12 hours thereafter. It may be extended to 24 hours at the discretion of the investigator.

Day 4 to Day 7: After an overnight fast from midnight, fluconazole will be administered in a dose of 800 mg on day 4 and 400 mg daily on Days 5-7 in the morning.

On Day 4, pharmacokinetic blood samples will be drawn for fluconazole estimation at the following times in relation to dosing:

-5 minutes, 15, 30, 45, 60, 75, 90, 120 min. 3, 4, 6, 8, 10, 12, 16, 20 hours.

Blood samples for determination of peak (4 hours) and trough (predose) plasma levels of fluconazole will be collected on Days 5 to 7 inclusive. Dosing on these days will be before breakfast is taken.

Vital signs (supine and standing pulse rate and blood pressure and oral temperature) will be recorded prior to dosing on Day 4 and at the following times thereafter:

1, 4, 8, 12, 24, 48 hours

12 lead ECGs will be recorded prior to dosing on Day 4 and at the following times thereafter:

24, 48 hours.

Fasting blood samples will be obtained for haematology, coagulation and clinical chemistry prior to dosing with fluconazole on Day 4 and at the following time points:

48 hours

A spot urine sample will be obtained for urinalysis prior to dosing with fluconazole on Day 4 and at the following time points:

48 hours

Days 8-11: Subjects will fast for 12 hours before dosing on Day 8. Water will be allowed ad libitum. Blood samples for determination of baseline plasma levels of fluconazole and F901318 blank and safety laboratory analyses (clinical chemistry, haematology and coagulation function) will be collected pre-dose on Day 8. F901318 (2 mg/kg IV for cohort 1 and up to 4 mg/kg IV for cohort 2) will be administered intravenously over 4 hours in the morning. Fluconazole will be administered orally on Day 8 at the same time as the start of the infusion. Blood samples for determination of plasma levels of fluconazole will be collected at the following time points after the dose of fluconazole:

15, 30, 45, 60, 75, 90 min, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 36, 48, 72 hours.

Blood samples for plasma concentrations of F901318 will be collected at the following times after the start of the infusion (assuming an infusion duration of 4 hours).

1, 2, 3, 4, 4.25, 4.5, 5, 6, 8, 10, 12, 16, 20, 24, 38, 48, 72 hours

Blood pressure, and pulse (lying and standing) and core temperature will be recorded at the following times on Day 8:

1. 2, 4, 6, 8, 12 and 24, 48, 72 hours following the start of dosing with F901318.

   Twelve lead ECGs will be recorded at 1, 4, 8, 12, 24, 48, 72 hours after dosing with F901318.

   Telemetry will be commenced 1 hour prior to dosing with F901318 and will continue for 12 hours thereafter. This monitoring may be extended to 24 hours at the discretion of the Principal Investigator.

   Adverse events and concomitant medications will be recorded throughout.

   Subjects will be discharged after all 72 hours measurements and observations have been completed, so long as they are fit to leave in the opinion of the Investigator.

   Post Study Visit: (visit 3) After discharge on Day 11, all subjects will return to the study centre on days 16-20 to complete a post study follow-up visit.

   Total blood loss for each subject in this part of the study will be 202 mL approximately.

   Part 2

   Treatment Period (Day -1 to Day 8; visit 3):

   Subjects will be admitted to the clinical unit in the afternoon of Day -1 and will remain on site until completion of the 72-hour post fluconazole and F901318 dose study-related procedures on Day 8. Admission procedures (Day -1) include a review of inclusion/exclusion criteria, weight, vital signs, test for drugs of abuse, alcohol and smoking and pregnancy where appropriate (must be negative) and a review of concomitant medication and adverse events. Blood (haematology, clinical chemistry and coagulation function) and urine (urinalysis) will be obtained for safety evaluations. Subjects will fast from midnight.

   Day 1: F901318 up to 4 mg/kg IV over 4 hours bid will be administered starting at time 0 and fluconazole 800 mg orally at time 0. A second dose of F901318 (up to 4 mg/kg IV over 4 hours) will be given starting at 12 hours post the morning dose. Water will be allowed ad libitum. Blood samples for determination of plasma levels of F901318 will be collected predose and at the following time points:
2. 4, 4.25, 4.5, 5, 6, 8, 10, 12 (just before second infusion), 16 (5 minutes before end of infusion) hours.

Pharmacokinetic blood samples will be drawn for fluconazole estimation pre-dose at the following times after dosing:

15, 30, 45, 60, 75, 90, 120 min. 3, 4, 6, 8, 10, 12, 16, 20 hours.

Blood pressure, and pulse (lying and standing), and oral temperature will be recorded at the following times on Day 1:

Prior to dosing, 1, 2, 4, 6, 8 and 12 hours following dosing.

Twelve lead ECGs will be recorded prior to dosing and 1, 4, 8, and 12 hours after dosing.

Telemetry will be set up 1 hour prior to dosing with F901318 and will continue for 12 hours thereafter. This monitoring may be extended to 24 hours at the discretion of the Principal Investigator.

Local tolerability will be determined prior to dosing with F901318 and at the end of each infusion.

Day 2 to Day 8: F901318 will be administered intravenously twice daily (7 doses of up to 2.5 mg/kg each infused over 4 hours) (Days 2 to 5).

Fluconazole will be administered after fasting from 12 midnight in a dose of 400 mg daily in the morning for 4 doses (Days 2 to 5).

Blood samples for determination of peak (4 hours) and trough (predose) plasma levels of fluconazole and F901318 (prior to start of infusion and 5 minutes before end of infusion) will be collected on Days 2 to 4 inclusive.

Vital signs (supine and standing pulse rate and blood pressure, core temperature and local tolerability) will be recorded prior to and at the end of each infusion on Days 2, 3 and 4

12 lead ECGs will be recorded prior to morning dosing on Days 2, 3, 4 and 5

Fasting blood samples will be obtained for haematology, coagulation and clinical chemistry prior to dosing with fluconazole on Days 2, 5 and on Day 8 (72 hours after the last doses of F901318 and fluconazole).

A spot urine sample will be obtained for urinalysis prior to dosing with fluconazole on Days 2, 5 and on Day 8 (72 hours after the last doses of F901318 and fluconazole).

On Day 5, pharmacokinetic blood samples will be drawn for F901318 estimation at the following times in relation to dosing:

-5 minutes, 2, 4, 4.25, 4.5, 5, 6, 8, 10, 12, 16, 20, 24, 36, 48, 72 hours.

On Day 5, pharmacokinetic blood samples will be drawn for fluconazole estimation at the following times in relation to dosing:

-5 minutes, 15, 30, 45, 60, 75, 90, 120 min. 3, 4, 6, 8, 10, 12, 16, 20, 24, 36, 48, 72 hours.

Vital signs and local tolerability will be obtained prior to dosing on Day 5 and at the end of the F901318 infusion.

Telemetry will be set up 1 hour prior to dosing with F901318 on Day 5 and will continue for 12 hours thereafter. This monitoring may be extended to 24 hours at the discretion of the Principal Investigator.

Day 8: An ophthalmology assessment will be performed. Subjects will be discharged from the Unit following collection of the final assessments and blood samples and completion of the ophthalmology assessment.

Adverse events and concomitant medications will be recorded throughout.

Post Study Visit (visit 4):

After discharge on Day 8, all subjects will return to the study centre on days 13-17 to complete a post study follow-up visit.

Total blood loss for each subject in this part of the study will be 224 mL approximately.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males and females of any ethnic origin aged between 18 and 45 years of age and weighing 50-100 kg inclusive.
2. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is acceptable).
3. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.

Exclusion Criteria:

1. Male and female subjects who are not willing to use appropriate contraception during the study and for three months thereafter.
2. Subjects who have received any prescribed systemic or topical medication within 14 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the dose administration (with the exception of vitamin/mineral supplements and paracetamol) unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
4. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety. For at least 2 weeks prior to dosing and until all blood samples and observations are completed on Day 18 +/- 2 (Part 1) or Day 15 +/- 2 (Part 2), subjects will not be allowed to eat any food or drink any beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family e.g. kale, broccoli, watercress, spring greens, kohlrabi, Brussels sprouts, mustard and charbroiled meats.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | 5 days
  Adverse events

SECONDARY OUTCOMES:
Pharmacokinetics area under concentration/time curve 0-t | 5 days
  Area under concentration time curve 0-t

CONTACTS AND LOCATIONS:
Overall Officials: A Stewart, Principal Investigator — Celerion Ltd
Locations (1):
- CELERION, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No